CLINICAL TRIAL: NCT03252587
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Efficacy and Safety of BMS-986165 in Subjects With Systemic Lupus Erythematosus
Brief Title: An Investigational Study to Evaluate BMS-986165 in Participants With Systemic Lupus Erythematosus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IM011-021; 2017-001203-79 (EudraCT Number)
Record Dates: First submitted 2017-08-15; First posted 2017-08-17 (Actual); Results first posted 2022-09-10 (Actual); Last update posted 2022-12-20 (Actual); Status verified 2022-11

CONDITIONS: Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — deucravacitinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- BMS-986165 Dose 1 oral administration (Experimental)
  Interventions: Drug: BMS-986165
- BMS-986165 Dose 2 oral administration (Experimental)
  Interventions: Drug: BMS-986165
- BMS-986165 Dose 3 oral administration (Experimental)
  Interventions: Drug: BMS-986165
- Placebo oral administration (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: BMS-986165 — Specified dose on specified days
  Arms: BMS-986165 Dose 1 oral administration; BMS-986165 Dose 2 oral administration; BMS-986165 Dose 3 oral administration
Other: Placebo — Specified dose on specified days
  Arms: Placebo oral administration

SUMMARY:
This study will investigate BMS-986165 to assess its effects in participants with systemic lupus erythematosus (SLE).

ELIGIBILITY:
Inclusion Criteria:

* Systemic lupus erythematosus (SLE) disease diagnosed ≥ 24 weeks before the screening visit
* Meets the Systemic Lupus International Collaborating Clinics (SLICC) classification criteria for SLE
* One of the following: elevated antinuclear antibodies (ANA) ≥ 1:80 or positive anti- double-stranded deoxyribonucleic acid (dsDNA) (positive includes indeterminate results) or positive anti-Smith (anti-Sm) as determined by the central laboratory
* Total Systemic Lupus Erythematosus Disease Activity Index 2000 (SLEDAI-2K) score ≥ 6 points and clinical SLEDAI-2K score ≥ 4 points with joint involvement and/or rash [score must be confirmed by Central Review Services (CRS)]
* Men and women must agree to follow specific methods of contraception, if applicable

Exclusion Criteria:

* Drug-induced SLE, certain other autoimmune diseases, and active, severe lupus nephritis
* SLE overlap syndromes such as scleroderma and mixed connective tissue disease
* Clinically significant abnormalities on chest x-ray or electrocardiogram (ECG)
* History of any significant drug allergy

Other protocol defined inclusion/exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 363 (Actual)
Dates: Start 2017-09-21 (Actual); Primary Completion 2021-06-29 (Actual); Study Completion 2021-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (189):
- United States (55):
  - Local Institution - 0178, Birmingham, Alabama
  - Little Rock Diagnostic Clinic, Little Rock, Arkansas
  - Local Institution - 0023, El Cajon, California
  - BioSolutions Clinical Research Center, La Mesa, California
  - Los Angeles County Hospital and University of Southern California Medical Center, Los Angeles, California
  - University of California at Irvine College of Medicine, Orange, California
  - Local Institution - 0227, Palm Desert, California
  - Millennium Clinical Trials - Thousand Oaks, Thousand Oaks, California
  - The Lundquist Institute at Harbor-UCLA Medical Center, Torrance, California
  - Inland Rheumatology Clinical Trials, Upland, California
  - Local Institution - 0034, Farmington, Connecticut
  - Local Institution - 0195, New Haven, Connecticut
  - Local Institution - 0010, Aventura, Florida
  - Local Institution - 0066, Brandon, Florida
  - Local Institution - 0214, Gainesville, Florida
  - Local Institution - 0233, Orlando, Florida
  - Local Institution - 0057, Ormond Beach, Florida
  - Local Institution - 0002, Tamarac, Florida
  - Local Institution - 0038, Tampa, Florida
  - BayCare Medical Group, Tampa, Florida
  - Local Institution - 0206, Atlanta, Georgia
  - Local Institution - 0022, Decatur, Georgia
  - Local Institution - 0083, Lawrenceville, Georgia
  - Arthritis Research and Treatment Center, Stockbridge, Georgia
  - Klein & Associates, Cumberland, Maryland
  - Klein and Associates, Hagerstown, Maryland
  - Advanced Rheumatology - Lansing, Lansing, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Local Institution - 0011, Brooklyn, New York
  - SUNY Downstate Health Science University, Brooklyn, New York
  - Local Institution - 0082, Lake Success, New York
  - Local Institution - 0109, New York, New York
  - Local Institution - 0232, New York, New York
  - Local Institution - 0119, Chapel Hill, North Carolina
  - Local Institution - 0026, Charlotte, North Carolina
  - Local Institution - 0180, Oklahoma City, Oklahoma
  - Local Institution - 0197, Oklahoma City, Oklahoma
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania
  - Local Institution - 0174, Wyomissing, Pennsylvania
  - Local Institution - 0190, Charleston, South Carolina
  - Local Institution - 0001, Jackson, Tennessee
  - University of Tennessee Health Science Center, Memphis, Tennessee
  - Local Institution - 0087, Austin, Texas
  - Local Institution - 0086, Austin, Texas
  - Pioneer Research Solutions, Cypress, Texas
  - Baylor Research Institute, Dallas, Texas
  - Local Institution - 0193, Dallas, Texas
  - Local Institution - 0204, Houston, Texas
  - Local Institution - 0061, Houston, Texas
  - Local Institution - 0047, Mesquite, Texas
  - Arthritis and Osteoporosis Center of South Texas, San Antonio, Texas
  - Local Institution - 0171, Chesapeake, Virginia
  - University of Washington, Seattle, Washington
  - Arthritis Northwest, PLLC, Spokane, Washington
- Argentina (10):
  - Local Institution - 0166, Caba, Buenos Aires
  - Local Institution - 0139, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - 0185, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - 0136, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - 0138, Ciudad Autonoma de Buenos Aires, Buenos Aires
  - Local Institution - 0152, Rosario, Santa Fe Province
  - Local Institution - 0097, San Miguel de Tucum, Tucumán Province
  - Local Institution - 0096, Córdoba
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Local Institution - 0137, Mendoza
- Australia (2):
  - Local Institution - 0241, Maroochydore, Queensland
  - Heidelberg Repatriation Hospital, Heidelberg West, Victoria
- Brazil (10):
  - Local Institution - 0130, Salvador, Estado de Bahia
  - Local Institution - 0129, Goiânia, Goiás
  - Santa Casa de Misericordia de Belo Horizonte, Belo Horizonte, Minas Gerais
  - Local Institution - 0125, Juiz de Fora, Minas Gerais
  - Local Institution - 0126, Curitiba, Paraná
  - Local Institution - 0128, Porto Alegre, Rio Grande do Sul
  - Hospital de Clinicas de Porto Alegre, Porto Alegre, São Paulo
  - Local Institution - 0151, São Bernardo do Campo, São Paulo
  - CITIPA - Centro de Imunoterapia de Ipanema, Rio de Janeiro
  - Local Institution - 0148, São Paulo
- Canada (4):
  - Local Institution - 0247, Calgary, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - McMaster University Medical Centre, Hamilton, Ontario
  - Local Institution - 0245, Toronto, Ontario
- Colombia (7):
  - Local Institution - 0098, Barranquilla
  - Local Institution - 0099, Barranquilla
  - Centro de Investigacion en Reumatologia y Especialidades Medicas (CIREEM), Bogotá
  - Medicity SAS, Bucaramanga
  - Local Institution - 0161, Cali
  - Local Institution - 0100, Chía
  - Local Institution - 0159, Zipaquirá
- Germany (3):
  - Allergie-Centrum-Charite Campus Charite Mitte Klinik fur Dermatologie Venerologie und Allergologi, Berlin
  - Klinik fur Nieren- und Hochdruckerkrankungen, Hanover
  - Universitatsmedizin der Johannes Gutenberg-Universitat Mainz - I. Medizinische Klinik und Poliklin, Mainz
- Hungary (4):
  - Del-pesti Centrumkorhaz - Orszagos Hematologiai es Infektologiai Intezet, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
  - Local Institution - 0035, Gyula
  - Local Institution - 0123, Szeged
- Israel (5):
  - Local Institution, Haifa
  - Local Institution, Jerusalem
  - Local Institution, Kfar Saba
  - Local Institution, Petah Tikva
  - Local Institution, Tel Litwinsky
- Japan (17):
  - Local Institution - 0117, Chiba, Chiba
  - Kameda Clinic, Kamogawa-shi, Chiba
  - Local Institution - 0177, Kitakyushu, Fukuoka
  - Hokkaido University Hospital, Sapporo, Hokkaido
  - Local Institution - 0141, Sapporo, Hokkaido
  - Tohoku University Hospital, Sendai, Miyagi
  - Tomishiro Central Hospital, Tomigusuku-shi, Okinawa
  - Dokkyo Medical University, Shimotsuga-gun, Tochigi
  - Local Institution - 0183, Shimotsuke, Tochigi
  - Local Institution - 0154, Chuo-ku, Tokyo
  - Local Institution - 0144, Itabashi-ku, Tokyo
  - Keio University Hospital, Shinjuku-Ku, Tokyo
  - Kanazawa University Hospital, Ishikawa
  - Local Institution - 0162, Tokyo
  - Showa University Hospital, Tokyo
  - National Hospital Organization Tokyo Medical Center, Tokyo
  - Local Institution - 0133, Tokyo
- Mexico (10):
  - Local Institution - 0163, León, Guanajuato
  - Local Institution - 0172, León, Guanajuato
  - Local Institution - 0135, Guadalajara, Jalisco
  - Local Institution - 0156, Zapopan, Jalisco
  - Juan Alberto Rodriguez Ruiz, Zapopan, Jalisco
  - Local Institution - 0173, Mexico City, Mexico City
  - Local Institution - 0140, Mexico City, Mexico City
  - Local Institution - 0134, Monterrey, Nuevo León
  - Local Institution - 0149, San Luis Potosí City
  - Faicic S. de R.L. de C.V., Veracruz
- Poland (23):
  - Local Institution - 0089, Bydgoszcz
  - Niepubliczny Zaklad Opieki Zdrowotnej BIF-MED S.C, Bytom
  - Centrum Kliniczno Badawcze J Brzezicki B Gornikiewicz Brzezicka Lekarze Spolka Partnerska, Elblag
  - Centrum Medyczne Pratia w Gdyni, Gdynia
  - Zespol Opieki Zdrowotnej w Konskich, Gmina Końskie
  - Silmedic Sp. z o.o., Katowice
  - Local Institution - 0182, Kościan
  - Local Institution - 0211, Krakow
  - Local Institution - 0222, Krakow
  - Centrum Medyczne ProMiMed, Krak
  - REUMED Sp. z o.o., Lublin
  - Medyczne Centrum Hetmanska - Poznan, Poznan
  - Solumed Centrum Medyczne, Poznan
  - Niepubliczny Specjalistyczny Zaklad Opieki Zdrowotnej Med-Polonia, Poznan
  - Local Institution - 0093, Sosnowiec
  - SANUS Szpital Specjalistyczny, Stalowa Wola
  - Local Institution - 0219, Warsaw
  - Local Institution - 0192, Warsaw
  - Local Institution - 0090, Warsaw
  - Centrum Medyczne AMED Warszawa Targowek, Warsaw
  - Local Institution - 0077, Wroclaw
  - Local Institution - 0184, Wroclaw
  - Local Institution - 0025, Wroclaw
- Romania (7):
  - Neomed Research, Brasov
  - Centrul Medical Sana, Bucharest
  - Spitalul Sfanta Maria, Bucharest
  - Spitalul Clinic Dr. Ioan Cantacuzino, Bucharest
  - Spitalul Clinic Judetean de Urgenta Cluj-Napoca, Cluj-Napoca
  - Spitalul Clinic Judeߥan de Urgenߡ Sfantul Apostol Andrei, Galati
  - Spitalul Judetean de Urgenta Valcea, Râmnicu Vâlcea
- Russia (15):
  - Kemerovo State Medical University, Kemerovo
  - Medical Center Maksimum Zdorovia, Kemerovo
  - Local Institution - 0210, Novosibirsk
  - Local Institution - 0006, Orenburg
  - State Healthcare Institution of the Republic of Karelia-Republican Hospital im.V.A.Baranova, Petrozavodsk
  - Clinical Rheumatological Hospital Number 25, Saint Petersburg
  - Local Institution - 0207, Saint Petersburg
  - Polyclinic of Private Security Personnel, Saint Petersburg
  - Local Institution - 0223, Saint Petersburg
  - Private Healthcare Institution Clinical Hospital, Smolensk
  - Tolyatti city clinical hospital ߵ, Tolyatti
  - Biomed, Vladimir
  - Local Institution - 0208, Yaroslavl
  - State Budgetary Healthcare Institution of the Yaroslavl Region Clinical Hospital No. 2, Yaroslavl
  - CjSC, Yekaterinburg
- South Korea (6):
  - Local Institution, Daegu
  - Local Institution, Daejeon
  - Local Institution - 0253, Gwangju
  - Local Institution, Incheon
  - Local Institution - 0054, Seoul
  - Local Institution - 0050, Suwon
- Spain (6):
  - Complejo Hospitalario Universitario A Coruna, A Coru
  - Hospital Universitari Vall dHebron, Barcelona
  - Hospital Regional Universitario de Malaga Hospital General, Málaga
  - Hospital de Merida, Mérida
  - Corporacio Sanitaria Parc Tauli, Sabadell
  - Local Institution - 0228, Seville
- Taiwan (5):
  - Local Institution, Changhua
  - Local Institution - 0114, Taichung
  - Local Institution - 0088, Taipei
  - Local Institution, Taipei
  - Local Institution, Taoyuan District

REFERENCES:
- [Derived] Mosca M, Arnaud L, Askanase A, Hobar C, Becker B, Singhal S, Banerjee S, Pomponi S, Choi J, Strand V. Deucravacitinib, an oral, selective, allosteric, tyrosine kinase 2 inhibitor, in patients with active SLE: efficacy on patient-reported outcomes in a phase II randomised trial. Lupus Sci Med. 2025 Jun 1;12(1):e001517. doi: 10.1136/lupus-2025-001517. PMID 40451616
- [Derived] Morand E, Pike M, Merrill JT, van Vollenhoven R, Werth VP, Hobar C, Delev N, Shah V, Sharkey B, Wegman T, Catlett I, Banerjee S, Singhal S. Deucravacitinib, a Tyrosine Kinase 2 Inhibitor, in Systemic Lupus Erythematosus: A Phase II, Randomized, Double-Blind, Placebo-Controlled Trial. Arthritis Rheumatol. 2023 Feb;75(2):242-252. doi: 10.1002/art.42391. Epub 2022 Nov 11. PMID 36369798
- [Derived] Hannon CW, McCourt C, Lima HC, Chen S, Bennett C. Interventions for cutaneous disease in systemic lupus erythematosus. Cochrane Database Syst Rev. 2021 Mar 9;3(3):CD007478. doi: 10.1002/14651858.CD007478.pub2. PMID 33687069
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo PO BID
- BMS-986165 3 mg: BMS-986165 3 mg PO BID
- BMS-986165 6 mg: BMS-986165 6 mg PO BID
- BMS-986165 12 mg: BMS-986165 12 mg PO QD
Period: Overall Study
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Started (Started = Randomized and treated) | 90 | 91 | 93 | 89
Completed (Completed = Completed treatment) | 66 | 71 | 76 | 62
Not Completed | 24 | 20 | 17 | 27
Not completed — Adverse Event | 3 | 8 | 6 | 12
Not completed — Lack of Efficacy | 7 | 2 | 2 | 4
Not completed — Lost to Follow-up | 2 | 0 | 0 | 2
Not completed — Pregnancy | 2 | 1 | 0 | 1
Not completed — Withdrawal by Subject | 8 | 4 | 4 | 4
Not completed — Other Reasons | 2 | 5 | 5 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg | Total
Number analyzed (Participants) | 90 | 91 | 93 | 89 | 363
Age, Continuous [Mean (Standard Deviation); unit: Years] | 40.1 (13.1) | 40.2 (11.9) | 40.9 (12.5) | 39.0 (10.6) | 40.1 (12.0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 80 | 85 | 88 | 81 | 334
  Male | 10 | 6 | 5 | 8 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 31 | 31 | 29 | 36 | 127
  Not Hispanic or Latino | 58 | 60 | 64 | 53 | 235
  Unknown or Not Reported | 1 | 0 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 4 | 3 | 5 | 2 | 14
  Asian | 10 | 9 | 15 | 10 | 44
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 6 | 10 | 8 | 9 | 33
  White | 60 | 62 | 55 | 57 | 234
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 10 | 7 | 10 | 11 | 38

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Meet Response Criteria for Systemic Lupus Erythematosus (SLE) Responder Index [SRI(4)] at Week 32
Description: SRI(4) responder is defined as a patient whose disease course fulfills all of the following:
  1. A 4-point or greater reduction from baseline in SLEDAI-2K score
  2. No new British Isles Lupus Assessment Group (BILAG) A (severe disease activity) and not more than 1 new BILAG B (moderate disease activity) organ domain grade
  3. No worsening from baseline in the Physician's Global Assessment of Disease Activity Scale by more than 0.3 points on a 3-point visual analog scale from no disease activity to severe disease activity
Time Frame: At week 32
Population: All Randomized Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 90 | 91 | 93 | 89
Participants | 31 | 53 | 46 | 40
Statistical Analysis 1: Comparison: Placebo vs BMS-986165 3 mg; BMS-986165 3 mg vs Placebo; Test type: Superiority; p = 0.0006, Regression, Logistic; 1-sided; Odds Ratio (OR) = 2.8, 95% CI 2-sided [1.5 to 5.1]
Statistical Analysis 2: Comparison: Placebo vs BMS-986165 6 mg; BMS-986165 6 mg vs Placebo; Test type: Superiority; p = 0.0210, Regression, Logistic; 1-sided; Odds Ratio (OR) = 1.9, 95% CI 2-sided [1.0 to 3.4]
Statistical Analysis 3: Comparison: Placebo vs BMS-986165 12 mg; BMS-986165 12 mg vs Placebo; Test type: Superiority; p = 0.0781, Regression, Logistic; 1-sided; Odds Ratio (OR) = 1.6, 95% CI 2-sided [0.8 to 2.9]

2. Secondary Outcome: Number of Participants Who Meet Response Criteria for Systemic Lupus Erythematosus (SLE) Responder Index [SRI(4)] at Week 48
Description: SRI(4) responder is defined as a patient whose disease course fulfills all of the following:
  1. A 4-point or greater reduction from baseline in SLEDAI-2K score
  2. No new British Isles Lupus Assessment Group (BILAG) A (severe disease activity) or not more than 1 new BILAG B (moderate disease activity) organ domain grade
  3. No worsening from baseline in the Physician's Global Assessment of Disease Activity Scale by more than 0.3 points on a 3-point visual analog scale from no disease activity to severe disease activity
Time Frame: At week 48
Population: All Randomized Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 90 | 91 | 93 | 89
Participants | 31 | 52 | 44 | 42
Statistical Analysis 1: Comparison: Placebo vs BMS-986165 3 mg; BMS-986165 3 mg vs Placebo; Test type: Superiority; p = 0.0011, Regression, Logistic; 1-sided; Odds Ratio (OR) = 2.6, 95% CI 2-sided [1.4 to 4.8]
Statistical Analysis 2: Comparison: Placebo vs BMS-986165 6 mg; BMS-986165 6 mg vs Placebo; Test type: Superiority; p = 0.0434, Regression, Logistic; 1-sided; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.9 to 3.1]
Statistical Analysis 3: Comparison: Placebo vs BMS-986165 12 mg; BMS-986165 12 mg vs Placebo; Test type: Superiority; p = 0.0439, Regression, Logistic; 1-sided; Odds Ratio (OR) = 1.7, 95% CI 2-sided [0.9 to 3.1]

3. Secondary Outcome: Number of Participants Who Achieve British Isles Lupus Assessment Group-Based Composite Lupus Assessment (BICLA) Response
Description: BICLA responder is defined as a patient whose disease course fulfills all of the following:
  1. Improvement in all organ systems with activity graded as BILAG-2004 A (severe disease activity) or B (moderate disease activity) at baseline
  2. No new organ system with activity graded as BILAG A; no more than 1 new organ system with activity graded as BILAG B
  3. No increase from baseline in Systemic Lupus Erythematosus SLEDAI-2K score (≤ 0 points for change from baseline score)
  4. No increase ≥ 10% in the Physician's Global Assessment of Disease Activity on a 3-point visual analog scale from no disease activity to severe disease activity
  5. No discontinuation of investigational product or use of restricted medications beyond the protocol allowed threshold before assessment
Time Frame: At week 48
Population: All Randomized Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 90 | 91 | 93 | 89
Participants | 23 | 43 | 33 | 32
Statistical Analysis 1: Comparison: Placebo vs BMS-986165 3 mg; BMS-986165 3 mg vs Placebo; Test type: Superiority; p = 0.0012, Regression, Logistic; 1-sided; Odds Ratio (OR) = 2.7, 95% CI 2-sided [1.4 to 5.1]
Statistical Analysis 2: Comparison: Placebo vs BMS-986165 6 mg; BMS-986165 6 mg vs Placebo; Test type: Superiority; p = 0.0795, Regression, Logistic; 1-sided; Odds Ratio (OR) = 1.6, 95% CI 2-sided [0.8 to 3.0]
Statistical Analysis 3: Comparison: Placebo vs BMS-986165 12 mg; BMS-986165 12 mg vs Placebo; Test type: Superiority; p = 0.0673, Regression, Logistic; 1-sided; Odds Ratio (OR) = 1.6, 95% CI 2-sided [0.9 to 3.2]

4. Secondary Outcome: Number of Participants Who Achieve Lupus Low Disease Activity State (LLDAS)
Description: LLDAS is defined as follows:
  1. SLEDAI-2K ≤ 4, with no activity in major organ systems (renal, central nervous system, cardiopulmonary, vasculitis, fever) and no hemolytic anemia or gastrointestinal activity measured as maintaining a D (no disease activity but suggests the system had previously been affected) or E (no current or previous disease activity) score in BILAG Gastrointestinal Body System
  2. No new lupus disease activity compared with the previous assessment measured as no new or worsening individual BILAG parameters
  3. Physician's Global Assessment of Disease Activity ≤ 1 on a 3-point visual analog scale from no disease activity to severe disease activity
  4. A current prednisolone (or equivalent) dose ≤ 7.5 mg daily
  5. Well-tolerated standard maintenance doses of immunosuppressive drugs and approved biological agents
Time Frame: At Week 48
Population: All Randomized Participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 90 | 91 | 93 | 89
Participants | 12 | 33 | 22 | 23
Statistical Analysis 1: Comparison: Placebo vs BMS-986165 3 mg; BMS-986165 3 mg vs Placebo; Test type: Superiority; p = 0.0002, Regression, Logistic; 1-sided; Odds Ratio (OR) = 4.0, 95% CI 2-sided [1.9 to 8.5]
Statistical Analysis 2: Comparison: Placebo vs BMS-986165 6 mg; BMS-986165 6 mg vs Placebo; Test type: Superiority; p = 0.0371, Regression, Logistic; 1-sided; Odds Ratio (OR) = 2.0, 95% CI 2-sided [0.9 to 4.5]
Statistical Analysis 3: Comparison: Placebo vs BMS-986165 12 mg; BMS-986165 12 mg vs Placebo; Test type: Superiority; p = 0.0168, Regression, Logistic; 1-sided; Odds Ratio (OR) = 2.3, 95% CI 2-sided [1.1 to 5.1]

5. Secondary Outcome: Number of Participants With a ≥50% Reduction in CLASI Activity Score in the Sub-group With Baseline CLASI Activity Score ≥10
Description: Number of participants with a Cutaneous Lupus Erythematosus Disease Area and Severity Index (CLASI) activity score ≥ 10 at baseline who achieve a CLASI response, defined as a decrease of ≥ 50% from baseline CLASI activity score (ranges from 0-70, where a higher score is associated with high disease activity). CLASI assesses by body surface area; points are given for presence of erythema, scale, hypertrophy, mucous membrane lesions, recent hair loss, and physician-observed alopecia
Time Frame: At week 48
Population: All Randomized Participants with Baseline CLASI Activity Score ≥ 10
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 24 | 23 | 25 | 29
Participants | 4 | 16 | 14 | 18
Statistical Analysis 1: Comparison: Placebo vs BMS-986165 3 mg; BMS-986165 3 mg vs Placebo; Test type: Superiority; p = 0.0006, Regression, Logistic; 1-sided; Odds Ratio (OR) = 10.5, 95% CI 2-sided [2.5 to 43.0]
Statistical Analysis 2: Comparison: Placebo vs BMS-986165 6 mg; BMS-986165 6 mg vs Placebo; Test type: Superiority; p = 0.0058, Regression, Logistic; 1-sided; Odds Ratio (OR) = 5.7, 95% CI 2-sided [1.5 to 22.0]
Statistical Analysis 3: Comparison: Placebo vs BMS-986165 12 mg; BMS-986165 12 mg vs Placebo; Test type: Superiority; p = 0.0009, Regression, Logistic; 1-sided; Odds Ratio (OR) = 8.2, 95% CI 2-sided [2.2 to 31.0]

6. Secondary Outcome: Change From Baseline in the 40-Joint Count
Description: Change from baseline in the following 40-joint count: phalangeal joints of the hand, second through fifth metacarpophalangeal joints of the hand, and individual metatarsophalangeal joints of the feet, Bilateral first metacarpophalangeal joints and shoulders. Each of 40 joints count is evaluated based upon the presence or absence of:
  1. Tender joint count (0 to 40)
  2. Swollen joint count (0 to 40)
  3. Tender and swollen joint count (0 to 40) A larger joint count indicates more severe disease.
Time Frame: Baseline and week 48
Population: All Randomized Participants
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 90 | 91 | 93 | 89
Units on a scale
  Tender: number analyzed (Participants) | 43 | 59 | 56 | 47
  Tender | -11.2 (8.0) | -12.2 (7.5) | -11.7 (9.5) | -12.3 (7.1)
  Swollen: number analyzed (Participants) | 43 | 59 | 56 | 47
  Swollen | -8.3 (6.9) | -8.5 (4.2) | -8.8 (7.2) | -9.9 (6.1)
  Tender + Swollen: number analyzed (Participants) | 43 | 59 | 56 | 47
  Tender + Swollen | -8.2 (6.7) | -8.2 (4.3) | -8.5 (7.0) | -9.7 (5.9)
Statistical Analysis 1: Comparison: Placebo vs BMS-986165 3 mg; Tender BMS-986165 3 mg vs Placebo; Test type: Superiority; p = 0.0131, Longitudinal Repeated Measures; Adjusted Mean Difference = -2.3, 95% CI 2-sided [-4.4 to -0.3], Standard Error of Mean 1.04
Statistical Analysis 2: Comparison: Placebo vs BMS-986165 6 mg; Tender BMS-986165 6 mg vs Placebo; Test type: Superiority; p = 0.4156, Longitudinal Repeated Measures; Adjusted Mean Difference = -0.2, 95% CI 2-sided [-2.3 to 1.8], Standard Error of Mean 1.04
Statistical Analysis 3: Comparison: Placebo vs BMS-986165 12 mg; Tender BMS-986165 12 mg vs Placebo; Test type: Superiority; p = 0.0151, Longitudinal Repeated Measures; Adjusted Mean Difference = -2.4, 95% CI 2-sided [-4.5 to -0.2], Standard Error of Mean 1.09
Statistical Analysis 4: Comparison: Placebo vs BMS-986165 3 mg; Swollen BMS-986165 3 mg vs Placebo; Test type: Superiority; p = 0.0029, Longitudinal Repeated Measures; Adjusted Mean Difference = -1.3, 95% CI 2-sided [-2.2 to -0.4], Standard Error of Mean 0.45
Statistical Analysis 5: Comparison: Placebo vs BMS-986165 6 mg; Swollen BMS-986165 6 mg vs Placebo; Test type: Superiority; p = 0.0516, Longitudinal Repeated Measures; Adjusted Mean Difference = -0.7, 95% CI 2-sided [-1.6 to 0.2], Standard Error of Mean 0.46
Statistical Analysis 6: Comparison: Placebo vs BMS-986165 12 mg; Swollen BMS-986165 12 mg vs Placebo; Test type: Superiority; p = 0.0298, Longitudinal Repeated Measures; Adjusted Mean Difference = -0.9, 95% CI 2-sided [-1.8 to 0.0], Standard Error of Mean 0.48
Statistical Analysis 7: Comparison: Placebo vs BMS-986165 3 mg; Tender + Swollen BMS-986165 3 mg vs Placebo; Test type: Superiority; p = 0.0010, Longitudinal Repeated Measures; Adjusted Mean Difference = -1.2, 95% CI 2-sided [-2.0 to -0.5], Standard Error of Mean 0.40
Statistical Analysis 8: Comparison: Placebo vs BMS-986165 6 mg; Tender + Swollen BMS-986165 6 mg vs Placebo; Test type: Superiority; p = 0.0343, Longitudinal Repeated Measures; Adjusted Mean Difference = -0.7, 95% CI 2-sided [-1.5 to 0.1], Standard Error of Mean 0.40
Statistical Analysis 9: Comparison: Placebo vs BMS-986165 12 mg; Tender + Swollen BMS-986165 12 mg vs Placebo; Test type: Superiority; p = 0.0050, Longitudinal Repeated Measures; Adjusted Mean Difference = -1.1, 95% CI 2-sided [-1.9 to -0.3], Standard Error of Mean 0.42

7. Secondary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Number of participants with any grade adverse events (AEs) and any grade serious adverse events (SAEs). An adverse event (AE) including SAEs is defined as any new untoward medical occurrence or worsening of a preexisting medical condition in participants that do not necessarily have causal relationship with treatment
Time Frame: From first dose to 30 days post last dose (Up to 52 weeks)
Population: All treated participants
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 90 | 91 | 93 | 89
Participants
  AEs | 79 | 85 | 81 | 75
  SAEs | 11 | 7 | 8 | 7

8. Secondary Outcome: Number of Participants With Laboratory Abnormalities in Specific Liver Tests
Description: Number of participants with laboratory abnormalities in specific liver tests based on US conventional units. The potential drug-induced liver injury is defined by the presence of all of the following:
  1. Alanine Aminotransferase (ALT) or Aspartate Aminotransferase (AST) elevation > 3× Upper Limit of Normal (ULN)
  2. Total bilirubin > 2× ULN, without initial findings of cholestasis (elevated serum alkaline phosphatase)
  3. No other immediately apparent possible causes of AST or AST elevation and hyperbilirubinemia, including, but not limited to, viral hepatitis, preexisting chronic or acute liver disease, or the administration of other drug(s) known to be hepatotoxic
Time Frame: From first dose to 30 days post last dose (Up to 52 weeks)
Population: All treated participants with evaluable measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 90 | 91 | 93 | 89
Participants
  ALT or AST > 3XULN: number analyzed (Participants) | 90 | 91 | 92 | 88
  ALT or AST > 3XULN | 2 | 5 | 3 | 2
  ALT or AST > 5XULN: number analyzed (Participants) | 90 | 91 | 92 | 88
  ALT or AST > 5XULN | 2 | 1 | 1 | 1
  Total Bilirubin > 2XULN: number analyzed (Participants) | 90 | 91 | 92 | 88
  Total Bilirubin > 2XULN | 0 | 0 | 0 | 0
  ALT or AST > 3XULN and Total Bilirubin > 2XULN on the same day: number analyzed (Participants) | 90 | 91 | 92 | 88
  ALT or AST > 3XULN and Total Bilirubin > 2XULN on the same day | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Participants With Abnormalities in Vital Signs
Description: Number of participants with abnormalities in vital signs including heart rate, systolic blood pressure, and diastolic blood pressure
Time Frame: From first dose to 30 days post last dose (Up to 52 weeks)
Population: All treated participants with evaluable measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 90 | 88 | 91 | 87
Participants
  Week 2: Heart Rate: Value > 100 and change from baseline > 30 | 0 | 0 | 0 | 0
  Week 2: Heart Rate: Value < 55 and change from baseline < -15 | 0 | 0 | 0 | 0
  Week 2: Systolic Blood Pressure: Value > 140 and change from baseline > 20 | 1 | 1 | 0 | 1
  Week 2: Systolic Blood Pressure: Value < 90 and change from baseline < -20 | 0 | 0 | 0 | 0
  Week 2: Diastolic Blood Pressure: Value > 90 and change from baseline > 10 | 0 | 0 | 1 | 1
  Week 2: Diastolic Blood Pressure: Value < 55 and change from baseline < -10 | 0 | 2 | 1 | 0
  Week 4: Heart Rate: Value > 100 and change from baseline > 30: number analyzed (Participants) | 89 | 86 | 91 | 84
  Week 4: Heart Rate: Value > 100 and change from baseline > 30 | 0 | 0 | 1 | 0
  Week 4: Heart Rate: Value < 55 and change from baseline < -15: number analyzed (Participants) | 89 | 86 | 91 | 84
  Week 4: Heart Rate: Value < 55 and change from baseline < -15 | 0 | 1 | 0 | 0
  Week 4: Systolic Blood Pressure: Value > 140 and change from baseline > 20: number analyzed (Participants) | 89 | 86 | 91 | 84
  Week 4: Systolic Blood Pressure: Value > 140 and change from baseline > 20 | 0 | 0 | 0 | 1
  Week 4: Systolic Blood Pressure: Value < 90 and change from baseline < -20: number analyzed (Participants) | 89 | 86 | 91 | 84
  Week 4: Systolic Blood Pressure: Value < 90 and change from baseline < -20 | 0 | 0 | 0 | 0
  Week 4: Diastolic Blood Pressure: Value > 90 and change from baseline > 10: number analyzed (Participants) | 89 | 86 | 91 | 84
  Week 4: Diastolic Blood Pressure: Value > 90 and change from baseline > 10 | 2 | 0 | 0 | 1
  Week 4: Diastolic Blood Pressure: Value < 55 and change from baseline < -10: number analyzed (Participants) | 89 | 86 | 91 | 84
  Week 4: Diastolic Blood Pressure: Value < 55 and change from baseline < -10 | 0 | 0 | 0 | 0
  Week 8: Heart Rate: Value > 100 and change from baseline > 30: number analyzed (Participants) | 87 | 86 | 88 | 81
  Week 8: Heart Rate: Value > 100 and change from baseline > 30 | 1 | 2 | 0 | 0
  Week 8: Heart Rate: Value < 55 and change from baseline < -15: number analyzed (Participants) | 87 | 86 | 88 | 81
  Week 8: Heart Rate: Value < 55 and change from baseline < -15 | 0 | 0 | 0 | 0
  Week 8: Systolic Blood Pressure: Value > 140 and change from baseline > 20: number analyzed (Participants) | 87 | 86 | 88 | 81
  Week 8: Systolic Blood Pressure: Value > 140 and change from baseline > 20 | 1 | 1 | 1 | 0
  Week 8: Systolic Blood Pressure: Value < 90 and change from baseline < -20: number analyzed (Participants) | 87 | 86 | 88 | 81
  Week 8: Systolic Blood Pressure: Value < 90 and change from baseline < -20 | 0 | 0 | 0 | 0
  Week 8: Diastolic Blood Pressure: Value > 90 and change from baseline > 10: number analyzed (Participants) | 87 | 86 | 88 | 81
  Week 8: Diastolic Blood Pressure: Value > 90 and change from baseline > 10 | 0 | 1 | 3 | 1
  Week 8: Diastolic Blood Pressure: Value < 55 and change from baseline < -10: number analyzed (Participants) | 87 | 86 | 88 | 81
  Week 8: Diastolic Blood Pressure: Value < 55 and change from baseline < -10 | 0 | 1 | 0 | 0
  Week 12: Heart Rate: Value > 100 and change from baseline > 30: number analyzed (Participants) | 79 | 86 | 84 | 75
  Week 12: Heart Rate: Value > 100 and change from baseline > 30 | 0 | 0 | 0 | 0
  Week 12: Heart Rate: Value < 55 and change from baseline < -15: number analyzed (Participants) | 79 | 86 | 84 | 75
  Week 12: Heart Rate: Value < 55 and change from baseline < -15 | 0 | 0 | 0 | 0
  Week 12: Systolic Blood Pressure: Value > 140 and change from baseline > 20: number analyzed (Participants) | 79 | 86 | 84 | 75
  Week 12: Systolic Blood Pressure: Value > 140 and change from baseline > 20 | 1 | 1 | 0 | 0
  Week 12: Systolic Blood Pressure: Value < 90 and change from baseline < -20: number analyzed (Participants) | 79 | 86 | 84 | 75
  Week 12: Systolic Blood Pressure: Value < 90 and change from baseline < -20 | 0 | 0 | 0 | 0
  Week 12: Diastolic Blood Pressure: Value > 90 and change from baseline > 10: number analyzed (Participants) | 79 | 86 | 84 | 75
  Week 12: Diastolic Blood Pressure: Value > 90 and change from baseline > 10 | 0 | 3 | 2 | 1
  Week 12: Diastolic Blood Pressure: Value < 55 and change from baseline < -10: number analyzed (Participants) | 79 | 86 | 84 | 75
  Week 12: Diastolic Blood Pressure: Value < 55 and change from baseline < -10 | 1 | 1 | 1 | 0
  Week 16: Heart Rate: Value > 100 and change from baseline > 30: number analyzed (Participants) | 79 | 79 | 83 | 76
  Week 16: Heart Rate: Value > 100 and change from baseline > 30 | 0 | 0 | 0 | 0
  Week 16: Heart Rate: Value < 55 and change from baseline < -15: number analyzed (Participants) | 79 | 79 | 83 | 76
  Week 16: Heart Rate: Value < 55 and change from baseline < -15 | 0 | 0 | 0 | 0
  Week 16: Systolic Blood Pressure: Value > 140 and change from baseline > 20: number analyzed (Participants) | 79 | 79 | 83 | 76
  Week 16: Systolic Blood Pressure: Value > 140 and change from baseline > 20 | 0 | 0 | 0 | 1
  Week 16: Systolic Blood Pressure: Value < 90 and change from baseline < -20: number analyzed (Participants) | 79 | 79 | 83 | 76
  Week 16: Systolic Blood Pressure: Value < 90 and change from baseline < -20 | 1 | 0 | 0 | 0
  Week 16: Diastolic Blood Pressure: Value > 90 and change from baseline > 10: number analyzed (Participants) | 79 | 79 | 83 | 76
  Week 16: Diastolic Blood Pressure: Value > 90 and change from baseline > 10 | 0 | 1 | 0 | 2
  Week 16: Diastolic Blood Pressure: Value < 55 and change from baseline < -10: number analyzed (Participants) | 79 | 79 | 83 | 76
  Week 16: Diastolic Blood Pressure: Value < 55 and change from baseline < -10 | 0 | 0 | 0 | 0
  Week 20: Heart Rate: Value > 100 and change from baseline > 30: number analyzed (Participants) | 77 | 81 | 82 | 74
  Week 20: Heart Rate: Value > 100 and change from baseline > 30 | 0 | 0 | 0 | 0
  Week 20: Heart Rate: Value < 55 and change from baseline < -15: number analyzed (Participants) | 77 | 81 | 82 | 74
  Week 20: Heart Rate: Value < 55 and change from baseline < -15 | 0 | 0 | 0 | 0
  Week 20: Systolic Blood Pressure: Value > 140 and change from baseline > 20: number analyzed (Participants) | 77 | 81 | 82 | 74
  Week 20: Systolic Blood Pressure: Value > 140 and change from baseline > 20 | 1 | 1 | 0 | 1
  Week 20: Systolic Blood Pressure: Value < 90 and change from baseline < -20: number analyzed (Participants) | 77 | 81 | 82 | 74
  Week 20: Systolic Blood Pressure: Value < 90 and change from baseline < -20 | 0 | 0 | 0 | 0
  Week 20: Diastolic Blood Pressure: Value > 90 and change from baseline > 10: number analyzed (Participants) | 77 | 81 | 82 | 74
  Week 20: Diastolic Blood Pressure: Value > 90 and change from baseline > 10 | 2 | 2 | 0 | 2
  Week 20: Diastolic Blood Pressure: Value < 55 and change from baseline < -10: number analyzed (Participants) | 77 | 81 | 82 | 74
  Week 20: Diastolic Blood Pressure: Value < 55 and change from baseline < -10 | 0 | 0 | 0 | 0
  Week 24: Heart Rate: Value > 100 and change from baseline > 30: number analyzed (Participants) | 69 | 78 | 80 | 69
  Week 24: Heart Rate: Value > 100 and change from baseline > 30 | 1 | 0 | 0 | 0
  Week 24: Heart Rate: Value < 55 and change from baseline < -15: number analyzed (Participants) | 69 | 78 | 80 | 69
  Week 24: Heart Rate: Value < 55 and change from baseline < -15 | 0 | 0 | 0 | 0
  Week 24: Systolic Blood Pressure: Value > 140 and change from baseline > 20: number analyzed (Participants) | 69 | 78 | 80 | 69
  Week 24: Systolic Blood Pressure: Value > 140 and change from baseline > 20 | 0 | 1 | 0 | 1
  Week 24: Systolic Blood Pressure: Value < 90 and change from baseline < -20: number analyzed (Participants) | 69 | 78 | 80 | 69
  Week 24: Systolic Blood Pressure: Value < 90 and change from baseline < -20 | 0 | 1 | 0 | 0
  Week 24: Diastolic Blood Pressure: Value > 90 and change from baseline > 10: number analyzed (Participants) | 69 | 78 | 80 | 69
  Week 24: Diastolic Blood Pressure: Value > 90 and change from baseline > 10 | 0 | 1 | 0 | 2
  Week 24: Diastolic Blood Pressure: Value < 55 and change from baseline < -10: number analyzed (Participants) | 69 | 78 | 80 | 69
  Week 24: Diastolic Blood Pressure: Value < 55 and change from baseline < -10 | 0 | 1 | 0 | 0
  Week 28: Heart Rate: Value > 100 and change from baseline > 30: number analyzed (Participants) | 68 | 76 | 80 | 66
  Week 28: Heart Rate: Value > 100 and change from baseline > 30 | 0 | 0 | 0 | 0
  Week 28: Heart Rate: Value < 55 and change from baseline < -15: number analyzed (Participants) | 68 | 76 | 80 | 66
  Week 28: Heart Rate: Value < 55 and change from baseline < -15 | 0 | 0 | 0 | 0
  Week 28: Systolic Blood Pressure: Value > 140 and change from baseline > 20: number analyzed (Participants) | 68 | 76 | 80 | 66
  Week 28: Systolic Blood Pressure: Value > 140 and change from baseline > 20 | 1 | 3 | 1 | 3
  Week 28: Systolic Blood Pressure: Value < 90 and change from baseline < -20: number analyzed (Participants) | 68 | 76 | 80 | 66
  Week 28: Systolic Blood Pressure: Value < 90 and change from baseline < -20 | 0 | 0 | 1 | 0
  Week 28: Diastolic Blood Pressure: Value > 90 and change from baseline > 10: number analyzed (Participants) | 68 | 76 | 80 | 66
  Week 28: Diastolic Blood Pressure: Value > 90 and change from baseline > 10 | 1 | 4 | 0 | 2
  Week 28: Diastolic Blood Pressure: Value < 55 and change from baseline < -10: number analyzed (Participants) | 68 | 76 | 80 | 66
  Week 28: Diastolic Blood Pressure: Value < 55 and change from baseline < -10 | 0 | 1 | 0 | 0
  Week 32: Heart Rate: Value > 100 and change from baseline > 30: number analyzed (Participants) | 67 | 75 | 78 | 63
  Week 32: Heart Rate: Value > 100 and change from baseline > 30 | 0 | 2 | 1 | 0
  Week 32: Heart Rate: Value < 55 and change from baseline < -15: number analyzed (Participants) | 67 | 75 | 78 | 63
  Week 32: Heart Rate: Value < 55 and change from baseline < -15 | 0 | 0 | 0 | 0
  Week 32: Systolic Blood Pressure: Value > 140 and change from baseline > 20: number analyzed (Participants) | 66 | 75 | 78 | 63
  Week 32: Systolic Blood Pressure: Value > 140 and change from baseline > 20 | 1 | 1 | 0 | 3
  Week 32: Systolic Blood Pressure: Value < 90 and change from baseline < -20: number analyzed (Participants) | 66 | 75 | 78 | 63
  Week 32: Systolic Blood Pressure: Value < 90 and change from baseline < -20 | 0 | 0 | 0 | 0
  Week 32: Diastolic Blood Pressure: Value > 90 and change from baseline > 10: number analyzed (Participants) | 66 | 75 | 78 | 63
  Week 32: Diastolic Blood Pressure: Value > 90 and change from baseline > 10 | 1 | 1 | 2 | 3
  Week 32: Diastolic Blood Pressure: Value < 55 and change from baseline < -10: number analyzed (Participants) | 66 | 75 | 78 | 63
  Week 32: Diastolic Blood Pressure: Value < 55 and change from baseline < -10 | 0 | 1 | 0 | 0
  Week 36: Heart Rate: Value > 100 and change from baseline > 30: number analyzed (Participants) | 65 | 72 | 79 | 61
  Week 36: Heart Rate: Value > 100 and change from baseline > 30 | 0 | 1 | 0 | 0
  Week 36: Heart Rate: Value < 55 and change from baseline < -15: number analyzed (Participants) | 65 | 72 | 79 | 61
  Week 36: Heart Rate: Value < 55 and change from baseline < -15 | 0 | 0 | 0 | 0
  Week 36: Systolic Blood Pressure: Value > 140 and change from baseline > 20: number analyzed (Participants) | 65 | 72 | 79 | 61
  Week 36: Systolic Blood Pressure: Value > 140 and change from baseline > 20 | 0 | 0 | 0 | 1
  Week 36: Systolic Blood Pressure: Value < 90 and change from baseline < -20: number analyzed (Participants) | 65 | 72 | 79 | 61
  Week 36: Systolic Blood Pressure: Value < 90 and change from baseline < -20 | 0 | 0 | 0 | 0
  Week 36: Diastolic Blood Pressure: Value > 90 and change from baseline > 10: number analyzed (Participants) | 65 | 72 | 79 | 61
  Week 36: Diastolic Blood Pressure: Value > 90 and change from baseline > 10 | 1 | 1 | 1 | 2
  Week 36: Diastolic Blood Pressure: Value < 55 and change from baseline < -10: number analyzed (Participants) | 65 | 72 | 79 | 61
  Week 36: Diastolic Blood Pressure: Value < 55 and change from baseline < -10 | 0 | 0 | 0 | 0
  Week 40: Heart Rate: Value > 100 and change from baseline > 30: number analyzed (Participants) | 63 | 73 | 78 | 62
  Week 40: Heart Rate: Value > 100 and change from baseline > 30 | 0 | 0 | 0 | 0
  Week 40: Heart Rate: Value < 55 and change from baseline < -15: number analyzed (Participants) | 63 | 73 | 78 | 62
  Week 40: Heart Rate: Value < 55 and change from baseline < -15 | 1 | 0 | 0 | 0
  Week 40: Systolic Blood Pressure: Value > 140 and change from baseline > 20: number analyzed (Participants) | 63 | 73 | 78 | 62
  Week 40: Systolic Blood Pressure: Value > 140 and change from baseline > 20 | 1 | 0 | 0 | 2
  Week 40: Systolic Blood Pressure: Value < 90 and change from baseline < -20: number analyzed (Participants) | 63 | 73 | 78 | 62
  Week 40: Systolic Blood Pressure: Value < 90 and change from baseline < -20 | 0 | 0 | 0 | 0
  Week 40: Diastolic Blood Pressure: Value > 90 and change from baseline > 10: number analyzed (Participants) | 63 | 73 | 78 | 62
  Week 40: Diastolic Blood Pressure: Value > 90 and change from baseline > 10 | 0 | 2 | 1 | 1
  Week 40: Diastolic Blood Pressure: Value < 55 and change from baseline < -10: number analyzed (Participants) | 63 | 73 | 78 | 62
  Week 40: Diastolic Blood Pressure: Value < 55 and change from baseline < -10 | 0 | 0 | 0 | 0
  Week 44: Heart Rate: Value > 100 and change from baseline > 30: number analyzed (Participants) | 66 | 72 | 73 | 62
  Week 44: Heart Rate: Value > 100 and change from baseline > 30 | 0 | 0 | 0 | 0
  Week 44: Heart Rate: Value < 55 and change from baseline < -15: number analyzed (Participants) | 66 | 72 | 73 | 62
  Week 44: Heart Rate: Value < 55 and change from baseline < -15 | 0 | 0 | 1 | 0
  Week 44: Systolic Blood Pressure: Value > 140 and change from baseline > 20: number analyzed (Participants) | 66 | 72 | 73 | 62
  Week 44: Systolic Blood Pressure: Value > 140 and change from baseline > 20 | 0 | 0 | 0 | 0
  Week 44: Systolic Blood Pressure: Value < 90 and change from baseline < -20: number analyzed (Participants) | 66 | 72 | 73 | 62
  Week 44: Systolic Blood Pressure: Value < 90 and change from baseline < -20 | 0 | 0 | 0 | 0
  Week 44: Diastolic Blood Pressure: Value > 90 and change from baseline > 10: number analyzed (Participants) | 66 | 72 | 73 | 62
  Week 44: Diastolic Blood Pressure: Value > 90 and change from baseline > 10 | 0 | 0 | 1 | 2
  Week 44: Diastolic Blood Pressure: Value < 55 and change from baseline < -10: number analyzed (Participants) | 66 | 72 | 73 | 62
  Week 44: Diastolic Blood Pressure: Value < 55 and change from baseline < -10 | 1 | 1 | 0 | 0
  Week 48: Heart Rate: Value > 100 and change from baseline > 30: number analyzed (Participants) | 64 | 69 | 75 | 61
  Week 48: Heart Rate: Value > 100 and change from baseline > 30 | 0 | 0 | 0 | 0
  Week 48: Heart Rate: Value < 55 and change from baseline < -15: number analyzed (Participants) | 64 | 69 | 75 | 61
  Week 48: Heart Rate: Value < 55 and change from baseline < -15 | 0 | 0 | 0 | 0
  Week 48: Systolic Blood Pressure: Value > 140 and change from baseline > 20: number analyzed (Participants) | 64 | 69 | 75 | 61
  Week 48: Systolic Blood Pressure: Value > 140 and change from baseline > 20 | 2 | 0 | 0 | 0
  Week 48: Systolic Blood Pressure: Value < 90 and change from baseline < -20: number analyzed (Participants) | 64 | 69 | 75 | 61
  Week 48: Systolic Blood Pressure: Value < 90 and change from baseline < -20 | 0 | 1 | 0 | 0
  Week 48: Diastolic Blood Pressure: Value > 90 and change from baseline > 10: number analyzed (Participants) | 64 | 69 | 75 | 61
  Week 48: Diastolic Blood Pressure: Value > 90 and change from baseline > 10 | 2 | 1 | 0 | 0
  Week 48: Diastolic Blood Pressure: Value < 55 and change from baseline < -10: number analyzed (Participants) | 64 | 69 | 75 | 61
  Week 48: Diastolic Blood Pressure: Value < 55 and change from baseline < -10 | 0 | 0 | 0 | 0
  Week 52: Heart Rate: Value > 100 and change from baseline > 30: number analyzed (Participants) | 8 | 11 | 12 | 14
  Week 52: Heart Rate: Value > 100 and change from baseline > 30 | 0 | 0 | 0 | 0
  Week 52: Heart Rate: Value < 55 and change from baseline < -15: number analyzed (Participants) | 8 | 11 | 12 | 14
  Week 52: Heart Rate: Value < 55 and change from baseline < -15 | 0 | 1 | 0 | 0
  Week 52: Systolic Blood Pressure: Value > 140 and change from baseline > 20: number analyzed (Participants) | 8 | 10 | 12 | 14
  Week 52: Systolic Blood Pressure: Value > 140 and change from baseline > 20 | 0 | 0 | 0 | 0
  Week 52: Systolic Blood Pressure: Value < 90 and change from baseline < -20: number analyzed (Participants) | 8 | 10 | 12 | 14
  Week 52: Systolic Blood Pressure: Value < 90 and change from baseline < -20 | 0 | 0 | 0 | 0
  Week 52: Diastolic Blood Pressure: Value > 90 and change from baseline > 10: number analyzed (Participants) | 8 | 10 | 12 | 14
  Week 52: Diastolic Blood Pressure: Value > 90 and change from baseline > 10 | 0 | 0 | 0 | 1
  Week 52: Diastolic Blood Pressure: Value < 55 and change from baseline < -10: number analyzed (Participants) | 8 | 10 | 12 | 14
  Week 52: Diastolic Blood Pressure: Value < 55 and change from baseline < -10 | 0 | 0 | 0 | 0

10. Secondary Outcome: Number of Participants With Abnormalities in Electrocardiograms (ECGs)
Description: Number of participants with abnormalities in electrocardiograms (ECGs) assessed by QTcF, PR interval, and QRS interval
Time Frame: From baseline to up to week 48
Population: All treated participants with evaluable measurements
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 89 | 90 | 92 | 89
Participants
  Baseline: QTcF 450 to < 480 | 9 | 3 | 6 | 5
  Baseline: QTcF 480 to < 500 | 1 | 1 | 0 | 0
  Baseline: QTcF >= 500 | 0 | 0 | 1 | 0
  Baseline: PR Interval >= 200 | 5 | 4 | 6 | 6
  Baseline: QRS Interval >=200 | 0 | 0 | 0 | 0
  Week 4: QTcF 450 to < 480: number analyzed (Participants) | 89 | 82 | 90 | 83
  Week 4: QTcF 450 to < 480 | 5 | 6 | 5 | 6
  Week 4: QTcF 480 to < 500: number analyzed (Participants) | 89 | 82 | 90 | 83
  Week 4: QTcF 480 to < 500 | 0 | 2 | 1 | 0
  Week4: QTcF >= 500: number analyzed (Participants) | 89 | 82 | 90 | 83
  Week4: QTcF >= 500 | 0 | 0 | 0 | 1
  Week 4: PR Interval >= 200: number analyzed (Participants) | 89 | 82 | 90 | 82
  Week 4: PR Interval >= 200 | 7 | 7 | 4 | 5
  Week 4: QRS Interval: >= 200: number analyzed (Participants) | 89 | 82 | 90 | 82
  Week 4: QRS Interval: >= 200 | 0 | 0 | 0 | 0
  Week 8: QTcF 450 to < 480: number analyzed (Participants) | 85 | 85 | 84 | 80
  Week 8: QTcF 450 to < 480 | 7 | 5 | 6 | 1
  Week 8: QTcF 480 to < 500: number analyzed (Participants) | 85 | 85 | 84 | 80
  Week 8: QTcF 480 to < 500 | 0 | 0 | 1 | 2
  Week 8: QTcF >=500: number analyzed (Participants) | 85 | 85 | 84 | 80
  Week 8: QTcF >=500 | 0 | 0 | 0 | 0
  Week 8: PR Interval >= 200: number analyzed (Participants) | 84 | 85 | 84 | 80
  Week 8: PR Interval >= 200 | 5 | 6 | 5 | 6
  Week 8 QRS Interval >=200: number analyzed (Participants) | 85 | 85 | 84 | 80
  Week 8 QRS Interval >=200 | 0 | 0 | 0 | 0
  Week 12: QTcF 450 to < 480: number analyzed (Participants) | 77 | 82 | 83 | 73
  Week 12: QTcF 450 to < 480 | 3 | 4 | 6 | 8
  Week 12: QTcF 480 to < 500: number analyzed (Participants) | 77 | 82 | 83 | 73
  Week 12: QTcF 480 to < 500 | 0 | 0 | 0 | 0
  Week 12: QTcF >= 500: number analyzed (Participants) | 77 | 82 | 83 | 73
  Week 12: QTcF >= 500 | 0 | 0 | 0 | 1
  Week 12: PR Interval >= 200: number analyzed (Participants) | 77 | 82 | 83 | 73
  Week 12: PR Interval >= 200 | 6 | 8 | 4 | 4
  Week 12: QRS Interval >=200: number analyzed (Participants) | 77 | 82 | 83 | 73
  Week 12: QRS Interval >=200 | 0 | 0 | 0 | 0
  Week 32: QTcF 450 to < 480: number analyzed (Participants) | 65 | 72 | 76 | 60
  Week 32: QTcF 450 to < 480 | 5 | 5 | 2 | 5
  Week 32: QTcF 480 to < 500: number analyzed (Participants) | 65 | 72 | 76 | 60
  Week 32: QTcF 480 to < 500 | 0 | 0 | 2 | 0
  Week 32: QTcF >=500: number analyzed (Participants) | 65 | 72 | 76 | 60
  Week 32: QTcF >=500 | 0 | 0 | 0 | 0
  Week 32: PR Interval >= 200: number analyzed (Participants) | 65 | 72 | 76 | 60
  Week 32: PR Interval >= 200 | 5 | 7 | 5 | 5
  Week 32: QRS Interval >= 200: number analyzed (Participants) | 65 | 72 | 76 | 60
  Week 32: QRS Interval >= 200 | 0 | 0 | 0 | 0
  Week 48: QTcF: 450 to < 480: number analyzed (Participants) | 63 | 67 | 72 | 58
  Week 48: QTcF: 450 to < 480 | 7 | 2 | 8 | 5
  Week 48: QTcF 480 to < 500: number analyzed (Participants) | 63 | 67 | 72 | 58
  Week 48: QTcF 480 to < 500 | 0 | 0 | 0 | 0
  Week 48: QTcF >=500: number analyzed (Participants) | 63 | 67 | 72 | 58
  Week 48: QTcF >=500 | 0 | 0 | 0 | 0
  Week 48: PR Interval: >= 200: number analyzed (Participants) | 63 | 67 | 72 | 58
  Week 48: PR Interval: >= 200 | 4 | 7 | 6 | 3
  Week 48: QRS Interval: >= 200: number analyzed (Participants) | 63 | 67 | 72 | 58
  Week 48: QRS Interval: >= 200 | 0 | 0 | 0 | 0

11. Secondary Outcome: BMS-986165 and Its Active Metabolite BMT-153261 Maximum Observed Plasma Concentration (Cmax)
Description: Maximum observed plasma concentration (Cmax) for the following treatments: BMS-986165 and its active metabolite BMT-153261. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
Time Frame: Pre-dose, 0.5, 2, 4, and 6 hours post dose on week 12
Population: All evaluable PK participants (all treated participants with available concentration-time data)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: NG/ML
Arm/Group | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 73 | 73 | 47
NG/ML
  BMS-986165: number analyzed (Participants) | 73 | 73 | 41
  BMS-986165 | 38.033 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 57.72 | 76.400 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 37.72 | 96.249 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 46.80
  Metabolite BMT-153261: number analyzed (Participants) | 68 | 72 | 47
  Metabolite BMT-153261 | 6.358 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 67.77 | 12.133 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 59.50 | 11.748 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 67.17

12. Secondary Outcome: BMS-986165 and Its Active Metabolite BMT-153261 Time of Maximum Observed Plasma Concentration (Tmax)
Description: Time of maximum observed plasma concentration (Tmax) for the following treatments: BMS-986165 and its active metabolite BMT-153261.
Time Frame: Pre-dose, 0.5, 2, 4, 6, and 10 hours post dose on week 12
Population: All evaluable PK participants (all treated participants with available concentration-time data)
Measure: Median (Full Range); unit: Hours
Arm/Group | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 73 | 73 | 47
Hours
  BMS-986165: number analyzed (Participants) | 73 | 73 | 41
  BMS-986165 | 2.0000 [0.467 to 6.000] | 2.0000 [0.500 to 7.533] | 2.0000 [0.500 to 5.100]
  Metabolite BMT-153261: number analyzed (Participants) | 68 | 72 | 47
  Metabolite BMT-153261 | 4.0000 [0.550 to 7.500] | 4.0000 [1.017 to 9.533] | 3.7330 [0.500 to 6.067]

13. Secondary Outcome: BMS-986165 and Its Active Metabolite BMT-153261 Trough Observed Plasma Concentration (Ctrough)
Description: Trough observed plasma concentration (Ctrough) for the following treatments: BMS-986165 and its active metabolite BMT-153261. Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported.
Time Frame: Pre-dose, 0.5, 2, 4, and 6 hours post dose on week 2, 4, 8, 12, 24, 32, and 48
Population: All evaluable PK participants (all treated participants with available concentration-time data)
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: NG/ML
Arm/Group | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 46 | 52 | 64
NG/ML
  BMS-986165 week 2: number analyzed (Participants) | 42 | 46 | 57
  BMS-986165 week 2 | 14.3737 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 60.790 | 29.2909 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 47.588 | 30.8135 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 70.340
  BMS-986165 week 4: number analyzed (Participants) | 36 | 42 | 64
  BMS-986165 week 4 | 14.6095 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 53.234 | 22.9170 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 51.043 | 20.1182 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 81.084
  BMS-986165 week 8: number analyzed (Participants) | 46 | 52 | 62
  BMS-986165 week 8 | 13.0328 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 69.792 | 12.9587 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 64.799 | 26.7961 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 67.090
  BMS-986165 week 12: number analyzed (Participants) | 43 | 46 | 64
  BMS-986165 week 12 | 10.7517 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 93.540 | 28.7751 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 47.282 | 22.1237 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 85.920
  BMS-986165 week 24: number analyzed (Participants) | 43 | 42 | 48
  BMS-986165 week 24 | 10.2546 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 66.763 | 13.9273 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 67.922 | 21.8720 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 78.559
  BMS-986165 week 32: number analyzed (Participants) | 38 | 41 | 41
  BMS-986165 week 32 | 8.5293 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 60.425 | 15.5285 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 61.704 | 24.5060 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 75.647
  BMS-986165 week 48: number analyzed (Participants) | 36 | 40 | 38
  BMS-986165 week 48 | 6.8493 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 70.206 | 21.7890 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 53.718 | 15.9576 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 102.367
  Metabolite BMT-153261 week 2: number analyzed (Participants) | 42 | 46 | 57
  Metabolite BMT-153261 week 2 | 4.2667 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 48.679 | 8.4841 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 54.717 | 8.7920 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 61.993
  Metabolite BMT-153261 week 4: number analyzed (Participants) | 36 | 42 | 64
  Metabolite BMT-153261 week 4 | 5.0886 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 56.764 | 7.7803 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 53.563 | 7.2703 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 70.461
  Metabolite BMT-153261 week 8: number analyzed (Participants) | 46 | 52 | 62
  Metabolite BMT-153261 week 8 | 4.1293 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 62.816 | 5.2290 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 71.924 | 8.1451 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 57.216
  Metabolite BMT-153261 week 12: number analyzed (Participants) | 43 | 46 | 64
  Metabolite BMT-153261 week 12 | 3.7325 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 96.323 | 9.3281 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 54.823 | 7.4071 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 82.009
  Metabolite BMT-153261 week 24: number analyzed (Participants) | 43 | 42 | 48
  Metabolite BMT-153261 week 24 | 3.3669 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 56.381 | 5.2229 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 71.104 | 6.6608 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 63.748
  Metabolite BMT-153261 week 32: number analyzed (Participants) | 38 | 41 | 41
  Metabolite BMT-153261 week 32 | 2.9759 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 55.379 | 5.2925 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 63.200 | 6.8734 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 77.329
  Metabolite BMT-153261 week 48: number analyzed (Participants) | 36 | 40 | 38
  Metabolite BMT-153261 week 48 | 2.8708 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 73.450 | 6.8838 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 58.302 | 5.8602 (NA) — Geometric coefficient of variation was not calculated and the arithmetic coefficient of variation (% CV) is being reported. %CV = 75.536

14. Secondary Outcome: Percent Change From Baseline in Interferon-Regulated Gene (IRG) Expression Levels
Description: Percent change from baseline in interferon-regulated gene (IRG) expression levels. IRG-high vs. IRG-low was determined using a 5-interferon (IFN) gene set during the sample collected at screening period. Baseline values are defined as the last measurement before the first dose.
Time Frame: From baseline to week 44
Population: All evaluable PD participants (all treated participants with at least one post-treatment measurement)
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 90 | 91 | 93 | 89
Percent Change from Baseline
  IFN High: number analyzed (Participants) | 65 | 76 | 73 | 69
  IFN High | -0.8130 (6.5323) | -39.7478 (13.0087) | -55.5691 (21.5313) | -47.5561 (12.2125)
  IFN Low: number analyzed (Participants) | 25 | 15 | 20 | 20
  IFN Low | 4.7381 (8.8696) | -18.0641 (27.0491) | -36.4510 (22.4759) | -41.7645 (26.1519)

15. Secondary Outcome: Percent Change From Baseline in Interferon-Regulated Gene (IRG) Expression Levels at Week 32
Description: as for outcome 14
Time Frame: From baseline to week 32
Population: All evaluable PD participants (all treated participants with at least one post-treatment measurement)
Measure: Mean (Standard Deviation); unit: Percent Change from Baseline
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 90 | 91 | 93 | 89
Percent Change from Baseline
  IFN High: number analyzed (Participants) | 65 | 76 | 73 | 69
  IFN High | -4.3993 (5.2234) | -40.7944 (13.5929) | -54.6988 (16.7734) | -61.0515 (13.8367)
  IFN Low: number analyzed (Participants) | 25 | 15 | 20 | 20
  IFN Low | -2.6555 (9.2649) | -27.4897 (20.0078) | -42.8107 (19.7669) | -42.9701 (23.8323)

16. Secondary Outcome: Percent Change From Baseline in Complement Proteins C3 and C4 Levels
Description: Percent change from baseline in complement proteins C3 and C4 levels. Baseline values are defined as the last measurement before the first dose.
Time Frame: From baseline to week 52
Population: All evaluable PD participants (all treated participants with at least one post-treatment measurement)
Measure: Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 8 | 10 | 12 | 14
Percent Change from Baseline
  C3 | 3.57 (12.225) | 5.33 (6.216) | 7.60 (5.315) | 14.74 (9.619)
  C4 | 84.52 (88.618) | 3.57 (7.146) | 24.96 (20.508) | 20.43 (12.767)

17. Secondary Outcome: Percent Change From Baseline in Complement (C3, C4) Levels at Week 32
Description: as for outcome 16
Time Frame: From baseline to week 32
Population: All evaluable PD participants (all treated participants with at least one post-treatment measurement)
Measure: Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 66 | 75 | 78 | 63
Percent Change from Baseline
  C3 | -0.58 (3.038) | 5.78 (3.161) | 12.42 (2.748) | 10.84 (2.896)
  C4 | -3.27 (3.297) | 12.32 (4.455) | 16.71 (5.012) | 25.13 (6.988)

18. Secondary Outcome: Percent Change From Baseline in Anti-Double-Stranded DNA (dsDNA) Antibody Levels
Description: Percent change from baseline in anti-double-stranded DNA (dsDNA) levels. Baseline values are defined as the last measurement before the first dose.
Time Frame: From baseline to week 52
Population: All evaluable PD participants (all treated participants with at least one post-treatment measurement)
Measure: Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 8 | 10 | 12 | 14
Percent Change from Baseline | 276.26 (316.713) | 16.51 (28.265) | -31.79 (10.209) | -19.32 (8.722)

19. Secondary Outcome: Percent Change From Baseline in Anti-Double-Stranded DNA (dsDNA) Antibody Levels at Week 32
Description: as for outcome 18
Time Frame: From baseline to week 32
Population: All evaluable PD participants (all treated participants with at least one post-treatment measurement)
Measure: Mean (Standard Error); unit: Percent Change from Baseline
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 64 | 75 | 77 | 63
Percent Change from Baseline | 21.36 (15.135) | -15.24 (4.910) | -11.31 (6.323) | -24.17 (4.781)

20. Secondary Outcome: Number of Participants With Global Systemic Lupus Erythematosus (SLE) Clinical Response Based on Interferon-Regulated Gene (IRG) Status
Description: Global systemic lupus erythematosus (SLE) clinical response in participants based on interferon-regulated gene (IRG) status (high versus low IRG signature). IRG-high vs. IRG-low was determined using a 5-interferon (IFN) gene set during the sample collected at screening period. SRI(4) responder is defined as a patient whose disease course fulfills all of the following:
  1. A 4-point or greater reduction from baseline in SLEDAI-2K score
  2. No new British Isles Lupus Assessment Group (BILAG) A (severe disease activity) or not more than 1 new BILAG B (moderate disease activity) organ domain grade
  3. No worsening from baseline in the Physician's Global Assessment of Disease Activity Scale by more than 0.3 points on a 3-point visual analog scale from no disease activity to severe disease activity
Time Frame: At week 32
Population: All randomized participants with SLE clinical response
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
Number analyzed (Participants) | 90 | 91 | 93 | 89
Participants
  IFN Low: number analyzed (Participants) | 25 | 15 | 20 | 20
  IFN Low | 10 | 7 | 11 | 5
  IFN High: number analyzed (Participants) | 65 | 76 | 73 | 69
  IFN High | 21 | 46 | 35 | 35

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) and Serious Adverse Events (SAEs) are collected from first dose to 30 days post last dose (Up to 52 weeks). Participants were assessed for All-cause mortality from their date of randomization to study completion (Up to 49 months)
Arm/Group | Placebo | BMS-986165 3 mg | BMS-986165 6 mg | BMS-986165 12 mg
All-Cause Mortality (participants affected / at risk) | 0/90 | 0/91 | 0/93 | 0/89
Serious Adverse Events (participants affected / at risk) | 11/90 | 7/91 | 8/93 | 7/89
Other Adverse Events (participants affected / at risk) | 52/90 | 56/91 | 60/93 | 45/89
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=90) | BMS-986165 3 mg (N=91) | BMS-986165 6 mg (N=93) | BMS-986165 12 mg (N=89)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Deficiency anaemia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 1
Scleritis (Eye disorders) | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 1 | 1 | 0
Generalised oedema (General disorders) | 1 | 0 | 0 | 0
Oedema peripheral (General disorders) | 0 | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 0 | 0 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 0 | 0 | 1
COVID-19 (Infections and infestations) | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 1 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1 | 0
Pyelonephritis chronic (Infections and infestations) | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Forearm fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Systemic lupus erythematosus (Musculoskeletal and connective tissue disorders) | 2 | 0 | 2 | 0
Invasive ductal breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Squamous cell carcinoma of the vagina (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Dysarthria (Nervous system disorders) | 1 | 0 | 0 | 0
Epilepsy (Nervous system disorders) | 1 | 0 | 0 | 0
Hemiparesis (Nervous system disorders) | 1 | 0 | 0 | 0
Optic neuritis (Nervous system disorders) | 0 | 0 | 1 | 0
Seizure (Nervous system disorders) | 0 | 1 | 0 | 0
Spinal cord disorder (Nervous system disorders) | 0 | 0 | 0 | 1
Abortion spontaneous incomplete (Pregnancy, puerperium and perinatal conditions) | 1 | 0 | 0 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 1
Uterine haemorrhage (Reproductive system and breast disorders) | 0 | 0 | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0
Hypertensive crisis (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=90) | BMS-986165 3 mg (N=91) | BMS-986165 6 mg (N=93) | BMS-986165 12 mg (N=89)
Diarrhoea (Gastrointestinal disorders) | 5 | 4 | 8 | 3
Nausea (Gastrointestinal disorders) | 8 | 6 | 5 | 4
Vomiting (Gastrointestinal disorders) | 6 | 3 | 4 | 1
Bronchitis (Infections and infestations) | 6 | 3 | 5 | 0
Cystitis (Infections and infestations) | 0 | 5 | 1 | 2
Nasopharyngitis (Infections and infestations) | 11 | 8 | 13 | 8
Oral herpes (Infections and infestations) | 0 | 4 | 4 | 5
Pharyngitis (Infections and infestations) | 2 | 7 | 5 | 2
Sinusitis (Infections and infestations) | 2 | 4 | 5 | 0
Upper respiratory tract infection (Infections and infestations) | 8 | 13 | 18 | 8
Urinary tract infection (Infections and infestations) | 3 | 10 | 6 | 6
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 5 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 8 | 2
Headache (Nervous system disorders) | 15 | 7 | 8 | 11
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 5 | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 4 | 3 | 8 | 7
Rash (Skin and subcutaneous tissue disorders) | 0 | 2 | 3 | 7
Hypertension (Vascular disorders) | 3 | 4 | 3 | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2020-04-15): https://cdn.clinicaltrials.gov/large-docs/87/NCT03252587/Prot_000.pdf
  • Statistical Analysis Plan (2021-12-20): https://cdn.clinicaltrials.gov/large-docs/87/NCT03252587/SAP_001.pdf